CLINICAL TRIAL: NCT03021629
Title: Comparison of Vitamin D Status and Vitamin D Receptor Polymorphisms in Patients With High Myopia and Primary Open-angle Glaucoma
Status: Completed | Type: Observational
Sponsor: Lv Yingjuan (Other)
Responsible Party: Sponsor-Investigator, Lv Yingjuan, Director, Tianjin Medical University Eye Hospital
Organization: Tianjin Medical University Eye Hospital (Other)
Other Study IDs: tjykdxykyy6
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Last update posted 2017-07-18 (Actual); Status verified 2017-07

CONDITIONS: Vitamin D Deficiency; Primary Open-angle Glaucoma; High Myopia; Vitamin D Receptor Polymorphisms
MeSH Terms: conditions — Vitamin D Deficiency; Glaucoma, Open-Angle

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- primary open-angle glaucoma patients: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay
  Interventions: Other: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay
- high myopia patients: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay
  Interventions: Other: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay
- age-matched people: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay
  Interventions: Other: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay

INTERVENTIONS:
Other: Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay
  Other Names: Vitamin D receptor polymorphic analysis was studied by polymerase chain reaction-restriction fragment length polymorphism technique

SUMMARY:
Vitamin D deficiency is known to be significantly associated with high myopia. This study investigated the vitamin D status in patients with high myopia and primary open-angle glaucoma, in order to understand the relationship between high myopia and the development of primary open-angle glaucoma.110 primary open-angle glaucoma patients, 110 high myopia patients and 110 age-matched people in the Han population were enrolled. Serum levels of 1a, 25-Dihydroxyvitamin D3 were measured by an enzyme-linked immuno-absorbent assay.Vitamin D receptor polymorphic analysis was studied by polymerase chain reaction-restriction fragment length polymorphism technique.

ELIGIBILITY:
Inclusion Criteria:

-primary open-angle glaucoma (1) intraocular pressure above 21 mmHg or more in each eye without therapy; (2) wide anterior chamber angle; (3)glaucomatous optic neuropathy (Glaucomatous optic nerve damage was defined as cup-to-disc ratio higher than 0.7 or focal loss of the nerve fiber layer (notch) associated with a consistent glaucomatous visual field defect in at least one eye;(4) visual field loss consistent with optic nerve damage and visual fields were performed by using standard automated perimetry in at least one eye.

c(with refractive error >6D) were recruited.

Exclusion Criteria:

* the presence of any secondary glaucoma with an exfoliation syndrome or a history of ocular trauma, high myopia, macular degeneration, other ocular diseases, and also a known history of systemic diseases and administration of vitamin D3 or other analog.

High myopia patients with ocular disease such as glaucoma, a history of administration of vitamin D3 or other analog or a history of retinopathy or connective tissue disorders associated with myopia, such as Stickler or Marfan syndromes, were not included.

Ages: 55 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary open-angle glaucoma patients, high myopia patients and age-matched people in the Han population
Sampling Method: Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2013-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Serum levels of 1a, 25-Dihydroxyvitamin D3 | 1 day visit

SECONDARY OUTCOMES:
gene polymorphisms of vitamin D receptor | 1 day visit

CONTACTS AND LOCATIONS:
Locations (1):
- Tianjin Medical University Eye Hospital, Tianjin, Tianjin Municipality, China